CLINICAL TRIAL: NCT01779154
Title: Eosinophilic Gastrointestinal Disorders Patient Registry
Status: Withdrawn | Type: Observational
Why Stopped: funding not available
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 136132
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Eosinophilic Esophagitis; Eosinophilic Gastritis; Eosinophilic Enteritis; Eosinophilic Colitis
Keywords: eosinophilic esophagitis; eosinophilic gastritis; eosinophilic enteritis; eosinophilic colitis
MeSH Terms: conditions — Eosinophilic Esophagitis; Eosinophilic enteropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- eosinophilic gastrointestinal disorders: Individuals with a diagnosis of EGID including: eosinophilic esophagitis, eosinophilic gastritis, eosinophilic enteritis, eosinophilic colitis

SUMMARY:
The Eosinophilic Gastrointestinal Disorders (EGIDS) Registry is a longitudinal study that does not involve medical interventions, but serves as a record of demographics, characteristics of disease and treatment, utilization patterns, quality improvement measures and clinical outcomes. The database is proposed so that epidemiologic research can be performed and current and accurate data can be obtained regarding practice patterns, age and gender distributions, efficacy of treatment, clinical outcomes and changes in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* male or female participants of any race or ethnicity
* age 0 to 21 years
* diagnosis of EGID including: eosinophilic esophagitis, eosinophilic gastritis, eosinophilic enteritis, eosinophilic colitis

Exclusion Criteria:

* hypereosinophilic syndrome
* non-eosinophilic gastrointestinal or allergic disorder

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals with a diagnosis of an eosinophilic gastrointestinal disorder
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2016-05 (Actual); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
To define characteristics of an eosinophilic gastrointestinal disorder population in a rural southern state | After 12 months of data collection
  To develop a database of patients with eosinophilic gastrointestinal disorders so that epidemiologic research can be performed and current data can be obtained regarding practice patterns, age and gender distributions, efficacy of treatment, clinical outcomes and changes in quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Robbie D Pesek, MD, Principal Investigator — University of Arkansas for Medical Sciences / Arkansas Children's Hospital Research Institute
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Pesek RD, Rettiganti M, O'Brien E, Beckwith S, Daniel C, Luo C, Scurlock AM, Chandler P, Levy RA, Perry TT, Kennedy JL, Chervinskiy S, Vonlanthen M, Casteel H, Fiedorek SC, Gibbons T, Jones SM. Effects of allergen sensitization on response to therapy in children with eosinophilic esophagitis. Ann Allergy Asthma Immunol. 2017 Aug;119(2):177-183. doi: 10.1016/j.anai.2017.06.006. Epub 2017 Jul 1. PMID 28676207